CLINICAL TRIAL: NCT07378878
Title: Comparison of Sevoflurane and Propofol Administration on Postoperative Cognitive Dysfunction in Spinal Surgery Using the Mini-Mental State Examination (MMSE)
Acronym: SEVO-PROP-MMSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Isak Lambas, Principal Investigator - Department of Anesthesiology and Intensive Therapy, Universitas Sumatera Utara, Universitas Sumatera Utara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 88/KEPK/USU/2025
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Condition / Focus: Postoperative Cognitive Dysfunction (POCD) Following Spinal Surgery
Keywords: Postoperative Cognitive Dysfunction; POCD; Spinal Surgery; Sevoflurane; Propofol; General Anesthesia; Cognitive Function
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned to either the sevoflurane or propofol group. Cognitive function is assessed at multiple time points postoperatively using the MMSE.
Who Masked: Outcomes Assessor
Masking Description: Participants are aware of the anesthesia type, but outcome assessors performing MMSE tests are blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane Group (Experimental): Inhalational anesthesia using sevoflurane. Dose and duration will follow standard anesthetic protocols for spinal surgery. Cognitive outcomes will be measured postoperatively using MMSE.
  Interventions: Drug: Sevoflurane Administration
- Propofol Group (Experimental): Patients in this group will receive general anesthesia using propofol during elective spinal surgery. Postoperative cognitive function will be assessed using the Mini-Mental State Examination (MMSE) at 6 hours, 24 hours, 3 days, and 7 days after surgery.
  Interventions: Drug: Propofol Administration

INTERVENTIONS:
Drug: Sevoflurane Administration — Inhalational anesthesia using sevoflurane. Dose and duration will follow standard anesthetic protocols for spinal surgery. Cognitive outcomes will be measured postoperatively using MMSE.
  Arms: Sevoflurane Group
Drug: Propofol Administration — Intravenous anesthesia using propofol. Dose and duration will follow standard anesthetic protocols for spinal surgery. Cognitive outcomes will be measured postoperatively using MMSE.
  Arms: Propofol Group

SUMMARY:
This study aims to compare the effects of two commonly used anesthetic agents, sevoflurane and propofol, on cognitive function after spinal surgery. Postoperative cognitive dysfunction (POCD) is a common complication following general anesthesia, particularly in complex procedures such as spinal surgery. The Mini-Mental State Examination (MMSE) will be used to assess cognitive function before surgery and at multiple time points after surgery (6 hours, 24 hours, 3 days, and 7 days).

Twenty patients undergoing elective spinal surgery will be randomly assigned to receive either sevoflurane or propofol anesthesia. Cognitive outcomes will be measured and compared between the two groups. The study will evaluate whether propofol offers better preservation of cognitive function compared to sevoflurane, which has been associated with oxidative stress and hippocampal dysfunction.

The results of this study will provide important information for anesthesiologists and surgical teams regarding the choice of anesthetic agents to minimize cognitive decline after spinal surgery, improving patient safety and postoperative recovery.

DETAILED DESCRIPTION:
Background:

Postoperative cognitive dysfunction (POCD) is a recognized complication following general anesthesia, particularly in major surgeries such as spinal procedures. POCD can affect memory, attention, and other cognitive domains, impacting patient recovery, quality of life, and independence after surgery. Sevoflurane, an inhalational anesthetic, has been associated with neurotoxic effects including oxidative stress and hippocampal dysfunction, which may contribute to POCD. Propofol, an intravenous anesthetic, exhibits antioxidative and anti-inflammatory properties, potentially offering neuroprotective effects.

Objective:

The primary objective of this study is to compare the incidence and severity of POCD in patients undergoing spinal surgery under sevoflurane versus propofol anesthesia, as assessed by the Mini-Mental State Examination (MMSE).

Methods:

This is a single-blind, randomized controlled trial involving 20 adult patients scheduled for elective spinal surgery at Universitas Sumatera Utara / RSUP H. Adam Malik Medan. Patients will be randomly allocated into two groups (n=10 per group) to receive either sevoflurane or propofol for general anesthesia.

Cognitive Assessment:

MMSE will be administered at the following time points:

Preoperatively (baseline)

6 hours postoperatively

24 hours postoperatively

3 days postoperatively

7 days postoperatively

Outcomes:

Primary Outcome: MMSE score change from baseline at each postoperative time point.

Secondary Outcomes: Incidence of mild or moderate POCD, defined according to MMSE decline; comparison of cognitive recovery trends between groups.

Statistical Analysis:

Descriptive statistics for demographic data.

Independent t-tests and chi-square tests to compare cognitive outcomes between groups.

Pearson correlation for analyzing associations between variables.

Significance threshold: p < 0.05.

Expected Results:

It is hypothesized that patients receiving propofol will demonstrate more stable MMSE scores postoperatively, whereas patients receiving sevoflurane may experience significant cognitive decline, particularly at 3 and 7 days after surgery.

Significance:

The study will provide evidence-based guidance for anesthetic selection in spinal surgery to minimize the risk of postoperative cognitive decline. This may improve patient recovery, satisfaction, and overall outcomes in surgical care.

Ethical Considerations:

The study has been approved by the Universitas Sumatera Utara Ethical Review Board (No. 88/KEPK/USU/2025). Informed consent will be obtained from all participants prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for elective spinal surgery.

Age between 18 and 65 years.

ASA (American Society of Anesthesiologists) physical status I-II.

Able to give informed consent.

Willing to participate in all cognitive assessments (MMSE) before and after surgery.

Exclusion Criteria:

History of neurological disorders (e.g., dementia, stroke, epilepsy).

Severe psychiatric disorders.

Known allergy or contraindication to sevoflurane or propofol.

History of drug or alcohol abuse.

Patients undergoing emergency spinal surgery.

Inability to understand or complete MMSE assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Change in Mini-Mental State Examination (MMSE) Score | Preoperatively (baseline), 6 hours, 24 hours, 3 days, and 7 days postoperatively
  Cognitive function of participants will be assessed using the Mini-Mental State Examination (MMSE) at multiple time points postoperatively. The change from baseline MMSE scores will be compared between the sevoflurane and propofol groups to evaluate the incidence and severity of postoperative cognitive dysfunction (POCD).

CONTACTS AND LOCATIONS:
Overall Officials: Isak Isak, MD, Principal Investigator — Department of Anesthesiology and Intensive Therapy, University of North Sumatra
Locations (1):
- RSUP H. Adam Malik Medan, Medan, North Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided